CLINICAL TRIAL: NCT06271759
Title: Psychological Effects of a Set of Essential Oils - A Randomized Interventional Trial
Brief Title: Psychological Effects of a Set of Essential Oils
Acronym: PSYFRAG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bucharest (Other)
Collaborators: IFF (International Flavors & Fragrances) (Unknown)
Responsible Party: Principal Investigator, Cezar Giosan, Associate Professor of Psychology, University of Bucharest
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PSYFRAG
Record Dates: First submitted 2024-02-14; First posted 2024-02-22 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Stress; Anxiety; Well-Being, Psychological; Mood
Keywords: Fragrances; Essential Oils; Well-being; Psychological effects; Anxiety; Stress; Depression
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Fragrance 1 Group (Experimental): At-home administration of one of the four active stimuli (fragrances), according to the following protocol:
  1. Participants will complete a series of psychological scales (pre-measurements), tapping into mood, affective states, well-being.
  2. Participants will inhale the fragranced stimulus for approximately 10 minutes.
  3. After the completion of step 2, participants will engage in a neutral activity for about 15 minutes.
  4. Participants will complete a series of psychological scales (post-measurements).
  5. Participants will repeat this protocol one week apart.
  Interventions: Other: Fragrance inhalation
- Fragrance 2 Group (Experimental): At-home administration of one of the four active stimuli (fragrances), according to the following protocol:
  1. Participants will complete a series of psychological scales (pre-measurements), tapping into mood, affective states, well-being.
  2. Participants will inhale the fragranced stimulus for approximately 10 minutes.
  3. After the completion of step 2, participants will engage in a neutral activity for about 15 minutes.
  4. Participants will complete a series of psychological scales (post-measurements).
  5. Participants will repeat this protocol one week apart.
  Interventions: Other: Fragrance inhalation
- Fragrance 3 Group (Experimental): At-home administration of one of the four active stimuli (fragrances), according to the following protocol:
  1. Participants will complete a series of psychological scales (pre-measurements), tapping into mood, affective states, well-being.
  2. Participants will inhale the fragranced stimulus for approximately 10 minutes.
  3. After the completion of step 2, participants will engage in a neutral activity for about 15 minutes.
  4. Participants will complete a series of psychological scales (post-measurements).
  5. Participants will repeat this protocol one week apart.
  Interventions: Other: Fragrance inhalation
- Fragrance 4 Group (Experimental): At-home administration of one of the four active stimuli (fragrances), according to the following protocol:
  1. Participants will complete a series of psychological scales (pre-measurements), tapping into mood, affective states, well-being.
  2. Participants will inhale the fragranced stimulus for approximately 10 minutes.
  3. After the completion of step 2, participants will engage in a neutral activity for about 15 minutes.
  4. Participants will complete a series of psychological scales (post-measurements).
  5. Participants will repeat this protocol one week apart.
  Interventions: Other: Fragrance inhalation
- No Fragrance Group (No Intervention): At-home administration of the neutral/no-odor stimulus, according to the following protocol:
  1. Participants will complete a series of psychological scales (pre-measurements), tapping into mood, affective states, well-being.
  2. Participants will inhale the non-fragranced stimulus for approximately 10 minutes.
  3. After the completion of step 2, participants will engage in a neutral activity for about 15 minutes.
  4. Participants will complete a series of psychological scales (post-measurements).
  5. Participants will repeat this protocol one week apart.

INTERVENTIONS:
Other: Fragrance inhalation — Inhalation of fragranced essential oils
  Arms: Fragrance 1 Group; Fragrance 2 Group; Fragrance 3 Group; Fragrance 4 Group

SUMMARY:
The goal of this clinical trial is to test the effectiveness of an intervention designed to improve wellness through aromatherapy. The main question it aims to answer is whether this intervention can deliver beneficial psychological effects on stress, anxiety and mood, as well as overall well-being.

Participants will receive a bottle with a no/neutral odor or an essential oil (or a blend of essential oils) for home administration and will be asked to complete a series of scales pre and post self-administration twice one week apart.

DETAILED DESCRIPTION:
The potential beneficial effects of a set of Essential Oils (EO) are being tested in the form of a Randomized Clinical Trial (RCT). There are five conditions: a control (receiving a neutral/no-odor stimulus) and four active groups (receiving one of the four EO).

The study is a within-subjects/between-subjects design with five arms and involves comparisons between pre-intervention and post-intervention between: (a) Initial psychological states of the participants, and (b) After inhalation of the stimuli. Participants will be randomly allocated to one of the five experimental arms.

For medium effect sizes assumed (f = 0.25), 5 groups and two measurements in time (pre and post stimulus administration) a minimum of 80 subjects total sample size is needed.

Affective states (relaxation, contentment, happiness, motivation, tension), as well as data on mood; depression, anxiety, and stress will be assessed.

Data about familiarity, pleasantness and intensity of the stimuli will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adults (at least 18 years old)

Exclusion Criteria:

* Allergies to Essential Oils
* Medical conditions that could have an effect on sense of smell

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Affective states - relaxation | Up to three months
  Changes in momentary affective states are assessed with a Visual Analogue Scale (VAS). VAS are 10-cm long analog scales, scored 0-100.
Affective states - contentment | Up to three months
  Changes in momentary affective states are assessed with a Visual Analogue Scale (VAS). VAS are 10-cm long analog scales, scored 0-100.
Affective states - happiness | Up to three months
  Changes in momentary affective states are assessed with a Visual Analogue Scale (VAS). VAS are 10-cm long analog scales, scored 0-100.
Affective states - stress | Up to three months
  Changes in momentary affective states are assessed with a Visual Analogue Scale (VAS). VAS are 10-cm long analog scales, scored 0-100.
Affective states - motivation | Up to three months
  Changes in momentary affective states are assessed with a Visual Analogue Scale (VAS). VAS are 10-cm long analog scales, scored 0-100.
Affective states - tension | Up to three months
  Changes in momentary affective states are assessed with a Visual Analogue Scale (VAS). VAS are 10-cm long analog scales, scored 0-100.
Emotional changes | Up to three months
  Changes in emotional patterns are assessed based on their intensity, one of the three components of emotional reactivity from the Multidimensional Emotion Questionnaire (MEQ). The questionnaire represents a reliable general measure of emotional experience, focusing on 10 discrete emotions (5 positive and 5 negative). Intensity is rated on a 5-Likert scale that ranges from 1 - Very low to 5 - Very high.

SECONDARY OUTCOMES:
General mental health - Depression | Up to three months
  Depressive symptoms are assessed with the Depression, Anxiety and Stress Scale (DASS-21).
General mental health - Anxiety | Up to three months
  Anxiety symptoms are assessed with the Depression, Anxiety and Stress Scale (DASS-21).
General mental health - Stress | Up to three months
  Stress is assessed with the Depression, Anxiety and Stress Scale (DASS-21).

CONTACTS AND LOCATIONS:
Overall Officials: Cezar Giosan, PhD, Principal Investigator — University of Bucharest
Locations (1):
- University of Bucharest, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No